CLINICAL TRIAL: NCT02078895
Title: Prospective Randomized Evaluation of Peri-Ureteral and Intradetrusor Injection of Botulinum Toxin Type A for the Treatment of Ureteral Stent Related Pain and Irritative Voiding Symptoms
Brief Title: Randomization of Botox for Stent Pain and Irritative Voiding Symptoms
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to low enrollment
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Jaime Landman, Department of Urology Chair, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-9702
Record Dates: First submitted 2014-02-26; First posted 2014-03-05 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Lower Urinary Tract Discomfort; Stent Pain
Keywords: Lower Urinary tract discomfort , ureteral stent pain
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botox (Experimental): The experimental group will include ureteral stent placement with three peri-ureteral injections of Botox A and fourteen site-specific intradetrusor injections of Botox A.
  Interventions: Drug: Botox
- Control (No Intervention): The control group will involve a ureteral stent placement with no injection.

INTERVENTIONS:
Drug: Botox — Peri-Ureteral and Intradetrusor Injection of Botulinum Toxin Type A
  Other Names: Botulinum Toxin Type A
  Arms: Botox

SUMMARY:
Botulinum toxin type A (Botox A) has shown great success in treating certain urologic conditions. A recent study has documented that Botox injected around the ureteral orifice (or place where the tube that connects the kidney to the bladder enters the bladder), during placement of a ureteral stent (small rubber tube that facilitate drainage of urine from the kidney to the bladder), resulted in a marked decline in the amount of stent pain experienced by patients. This finding was quite remarkable as stents are commonly used in many Urologic conditions, and these stents produce a remarkable degree of patient discomfort. Despite the great improvement in pain reduction, the irritative voiding symptoms [frequent need to void, urgency, burning with urination (dysuria) or nighttime voiding (nocturia)] were not ameliorated by the Botox injections in the ureteral orifice. However, it has already been well documented that in other clinical settings, administrations of Botox into the bladder muscle, has been shown to reduce these irritative symptoms.

The objective of the study is to determine if pain and irritative lower urinary tract symptoms related to ureteral stent placement will improve after the injection of Botox around the ureteral orifice and in the bladder itself.

DETAILED DESCRIPTION:
The objective of this prospective randomized single blinded controlled pilot study for patients undergoing unilateral ureteral stent insertion for benign urologic conditions is to determine if pain and irritative lower urinary tract symptoms (frequency, urgency, dysuria, nocturia) related to ureteral stent placement will improve after the injection of intradetrusor Botox (BTX) A.

The effects of BTX have been used for a number of medicinal purposes, including reducing wrinkles, migraine headaches, and excessive sweating. The use of BTX in urology and, more specifically, the lower urinary tract, is increasing. Botox is currently actively being used as a treatment strategy for use in Urologic conditions including neurogenic and non-neurogenic overactive bladder (OAB), detrusor sphincter dyssynergia, interstitial cystitis, urinary retention, and prostate disorders.

BTX serotypes. The seven distinct serotypes of BTX are designated A, B, C1, E, F, and G; BTX-A (Botox [Allergan, Inc., Irvine, Calif] and Dysport [Ipsen, Inc., Europe]) and BTX-B (Myobloc (Solstice Neurosciences, Inc., Malvern, Pa) are available commercially. Each serotype of botulinum toxin works by inhibiting the release of neurotransmitters, most notably acetylcholine, from the presynaptic neuromuscular junction (2). The result is inhibition of muscular contractions and paralysis.

In August 2011, the FDA recently approved the use of Botox injections for urinary incontinence secondary to neurogenic overactive bladder, a condition defined as unihibited bladder contractions causing voiding and creating symptoms of urinary frequency. The cause of the neurogenic overactive bladder in the patients studied was spinal cord injury and multiple sclerosis. Numerous prospective clinical trials have demonstrated a statistically significant difference of symptoms in patients receiving Botox injections into the overactive detrusor muscle compared to placebo groups. Botox injections were found to effectively relieve urinary incontinence and urinary frequency for a nine-month duration.

As part of standard clinical care, intravesical injection of Botox is currently used to ameliorate voiding symptoms in conditions where patients experience severe irritative symptoms and is currently seeking FDA approval for the treatment of overactive bladder in patients without a neurologic etiology. As a follow up study, we will evaluate the efficacy of combined periureteral and intravesical Botox injection for reduction of pain and irritative voiding

This is a prospective randomized single blinded controlled study for patients undergoing unilateral ureteral stent insertion for a benign urologic conditions is to determine if pain and irritative lower urinary tract symptoms (frequency, urgency, dysuria, nocturia) related to ureteral stent placement will improve after the injection of intradetrusor Botox A.

Study in detail:

All patients will be informed regarding the content of the study and informed consent will be obtained. Patients who require stent placement will be screened based on their past medical history and will be included in the study if they do not fit any of the exclusion criteria. The participation in the study will require 3 visits in addition to pre-op visit when the consent will be obtained: stent placement, stent removal, and 2 week post-op follow up. Patients will only have one pre-operative visit prior to ureteral stent placement. Patients will be randomized to one of two groups, experimental and placebo. The experimental group will include ureteral stent placement with three peri-ureteral injections of Botox A and fourteen site-specific intradetrusor injections of Botox A. The placebo group will involve a ureteral stent placement with no injection. Based on a randomization sequence from an electronic randomizer, patients will be placed in either Botox injection group or placebo (no injection) group. Patients will be consented at the pre-operative visit, which is usually up to seven days prior to the procedure. After informed consent is obtained, patients will be asked to complete a visual analog pain scale and a ureteral stent symptom questionnaire which can either be turned in during the pre-operative visit or alternatively, if the patient prefers to review the study prior to deciding to participate, can be turned in during the day of stent placement in the pre-operative area at UC Irvine Douglas Hospital before the procedure start time, giving the patient ample time to consider study participation. Baseline post-void residual will also be taken at the pre-operative visit. All stents will be inserted in a retrograde fashion as per standard of care. As standard of care, retrograde contrast injection following the procedure will be done to assess ureteral and renal anatomy. Jaime Landman, MD., and Gamal Ghoniem, MD., will be administering all Botox injections. Three 1mL Botox A injections (10U/mL) will be placed medial, lateral, and inferior to the ureteral orifice. Fourteen 1mL injections (5U/mL) will be placed into the detrusor muscle: three injections at the trigone avoiding the bladder neck, away from the peri-ureteral injections (10U/mL), and eleven injections distributed evenly across the remainder of the bladder. A total of 100 units (1 vial) of Botox A will be used per patient. 100 units of Botox A will be diluted with 10cc's of 0.9% PFNS, 3 cc's will be drawn for the peri-ureteral injections (30 units), then 7 ccs of 0.9% PFNS will be added to the vial to bring to 14cc's. The rest of the Botox A (70u) will be injected into the detrusor muscle.

Procedures will be planned for day surgeries and will be given one pre-operative dose of Kefzol for urinary tract infection prophylaxis as standard of care to all patients. The patient will subsequently be evaluated one hour after the procedure in the recovery room with a visual analog pain scale only. Subsequently, two post-operative evaluations will occur: On the day of stent removal, usually post-operative days (POD) 3 - 9, and POD 14 follow up, The patient will also be assessed during the second follow-up evaluation on POD's 3 - 9 for the possibility of urinary tract infection or urinary retention. A post-void residual will be taken during the 2 week follow-up to assess for urinary retention. On POD 14 visit, a USSQ, medication diary, visual pain analog scale will be collected from the patient. Post-operative evaluation will consist of a visual analog pain scale and a ureteral stent symptom questionnaire (USSQ) to assess pain, lower urinary tract symptoms, and quality of life. In addition, a narcotic diary will be kept by patients to determine the quantity and duration of oral narcotic required during the time the stent is in place. The narcotic diary is important in the study to assess the pain the patient is experiencing in addition to the visual pain analog scale that will be used. A standardized post-operative pain regimen will include Percocet (5mg Oxycodone/325mg Acetominophen) 1 - 2 tablets prn every 4 hours. Pain regimen of Percocet is standard of care and will not be used specifically for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring unilateral ureteral stent insertion
* Age > 18
* Renal/ureteral stones (single or multiple)
* Ureteral strictures
* Surveillance ureterscopy
* Willing and able to consent
* Willing and able to complete study questionnaires/diaries
* Willing to use CIC to empty the bladder at any time after study treatment if it is determined to be necessary by the investigator

Exclusion Criteria:

* History of malignancy
* Patients on medical therapy for benign prostatic hyperplasia (alpha blocker and/or 5alpha reductase inhibitor)
* Patients taking muscarinic-receptor antagonists (Ex. detrol, ditropan etc.)
* Patients who have an interstim sacral neuromodulator
* History of urinary retention
* Neurogenic or non-neurogenic detrusor overactivity
* Pregnancy
* Solitary kidney
* Insulin dependent Diabetes Mellitus (Uncontrolled Diabetes (HbA1c > 8))
* Neuropathy
* History of transplant kidney
* History of narcotic abuse or chronic pain
* Anatomic bladder/ureteral abnormality
* Previous cystectomy/urinary diversion
* Conditions necessitating bilateral ureteral stents
* History of Interstitial cystitis
* Patients with a post-void residual volume of > 100ml
* Patients with history of urinary retention
* Patients with active urinary tract infection
* Patients with history of chronic urinary tract infections
* Patients with concomitant use of any botulinum toxin within 3 months or any urological use of botulinum toxin in the past
* Patients with active genital infection, other than genital warts, either concurrently or within 4 weeks prior to screening
* Patients with concurrent or previously uninvestigated hematuria within 6 months prior to screening. -Patients with investigated hematuria may have entered the study if urological/renal pathology had been ruled out to the satisfaction of the investigator
* Patients with hemophilia, or other clotting factor deficiencies, or disorders that cause bleeding diathesis Patients with a known allergy or sensitivity to any botulinum toxin preparation (including study medication preparation), anesthetics, or antibiotics used during the study
* Patients with any medical condition that may have put them at increased risk with exposure to Botox including diagnosed myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in Lower Urinary Tract Discomfort between pre-operative visit date and the stent removal date and two week follow up. | At pre-operative visit (average of 7 days before stent placement), stent removal date (3-9 days after stent placement), and 2 week follow up (2 weeks after stent placement)
  Lower urinary tract symptoms (frequency, urgency, nocturia, dysuria) - Ureteral Stent Symptom Questionnaire (USSQ). The USSQ has different sections that pertain to different domains of a patient's life. Therefore, a total score from each section will be measured individually as described by Joshi et al (15). The different domains of the USSQ include urinary symptoms, body pain, general health, work performance, sexual matters. The total scores from each of these sections will be compared individually. In addition, the total score for the entire questionnaire will also be assessed.

SECONDARY OUTCOMES:
Post-operative pain | At pre-operative visit (average of 7 days before stent placement), stent removal date (3-9 days after stent placement), and 2 week follow up (2 weeks after stent placement)
  Post-operative pain - visual analog scale (VAS).
Post-surgical analgesic requirements | post-operative to follow up day (2 weeks)
  Post-surgical analgesic requirements: Oral opiates/-patients to keep written record (number/duration
  -# of days)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Landman, MD, Principal Investigator — University of California, Irvine Department of Urology
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta M, Patel T, Xavier K, Maruffo F, Lehman D, Walsh R, Landman J. Prospective randomized evaluation of periureteral botulinum toxin type A injection for ureteral stent pain reduction. J Urol. 2010 Feb;183(2):598-602. doi: 10.1016/j.juro.2009.10.021. Epub 2009 Dec 16. PMID 20018320
- [Background] Brin MF. Botulinum toxin: chemistry, pharmacology, toxicity, and immunology. Muscle Nerve Suppl. 1997;6:S146-68. PMID 9826987
- [Background] Herschorn S, Gajewski J, Ethans K, Corcos J, Carlson K, Bailly G, Bard R, Valiquette L, Baverstock R, Carr L, Radomski S. Efficacy of botulinum toxin A injection for neurogenic detrusor overactivity and urinary incontinence: a randomized, double-blind trial. J Urol. 2011 Jun;185(6):2229-35. doi: 10.1016/j.juro.2011.02.004. Epub 2011 Apr 16. PMID 21497851
- [Background] Kalsi V, Apostolidis A, Gonzales G, Elneil S, Dasgupta P, Fowler CJ. Early effect on the overactive bladder symptoms following botulinum neurotoxin type A injections for detrusor overactivity. Eur Urol. 2008 Jul;54(1):181-7. doi: 10.1016/j.eururo.2007.12.029. Epub 2007 Dec 26. PMID 18191323
- [Background] Schmid DM, Sauermann P, Werner M, Schuessler B, Blick N, Muentener M, Strebel RT, Perucchini D, Scheiner D, Schaer G, John H, Reitz A, Hauri D, Schurch B. Experience with 100 cases treated with botulinum-A toxin injections in the detrusor muscle for idiopathic overactive bladder syndrome refractory to anticholinergics. J Urol. 2006 Jul;176(1):177-85. doi: 10.1016/S0022-5347(06)00590-8. PMID 16753396
- [Background] Rapp DE, Lucioni A, Katz EE, O'Connor RC, Gerber GS, Bales GT. Use of botulinum-A toxin for the treatment of refractory overactive bladder symptoms: an initial experience. Urology. 2004 Jun;63(6):1071-5. doi: 10.1016/j.urology.2004.01.041. PMID 15183952
- [Background] Dykstra D, Enriquez A, Valley M. Treatment of overactive bladder with botulinum toxin type B: a pilot study. Int Urogynecol J Pelvic Floor Dysfunct. 2003 Dec;14(6):424-6. doi: 10.1007/s00192-003-1099-3. Epub 2003 Nov 25. PMID 14677005
- [Background] Ghei M, Maraj BH, Miller R, Nathan S, O'Sullivan C, Fowler CJ, Shah PJ, Malone-Lee J. Effects of botulinum toxin B on refractory detrusor overactivity: a randomized, double-blind, placebo controlled, crossover trial. J Urol. 2005 Nov;174(5):1873-7; discussion 1877. doi: 10.1097/01.ju.0000177477.83991.88. PMID 16217327
- [Background] Schurch B, Stohrer M, Kramer G, Schmid DM, Gaul G, Hauri D. Botulinum-A toxin for treating detrusor hyperreflexia in spinal cord injured patients: a new alternative to anticholinergic drugs? Preliminary results. J Urol. 2000 Sep;164(3 Pt 1):692-7. doi: 10.1097/00005392-200009010-00018. PMID 10953127
- [Background] Reitz A, Stohrer M, Kramer G, Del Popolo G, Chartier-Kastler E, Pannek J, Burgdorfer H, Gocking K, Madersbacher H, Schumacher S, Richter R, von Tobel J, Schurch B. European experience of 200 cases treated with botulinum-A toxin injections into the detrusor muscle for urinary incontinence due to neurogenic detrusor overactivity. Eur Urol. 2004 Apr;45(4):510-5. doi: 10.1016/j.eururo.2003.12.004. PMID 15041117
- [Background] Staskin DR, Dmochowski RR, Sand PK, Macdiarmid SA, Caramelli KE, Thomas H, Hoel G. Efficacy and safety of oxybutynin chloride topical gel for overactive bladder: a randomized, double-blind, placebo controlled, multicenter study. J Urol. 2009 Apr;181(4):1764-72. doi: 10.1016/j.juro.2008.11.125. Epub 2009 Feb 23. PMID 19233423
- [Background] Duvdevani M, Chew BH, Denstedt JD. Minimizing symptoms in patients with ureteric stents. Curr Opin Urol. 2006 Mar;16(2):77-82. doi: 10.1097/01.mou.0000193375.29942.0f. PMID 16479208
- [Background] Beiko DT, Knudsen BE, Denstedt JD. Advances in ureteral stent design. J Endourol. 2003 May;17(4):195-9. doi: 10.1089/089277903765444294. PMID 12816579
- [Background] Chew BH, Duvdevani M, Denstedt JD. New developments in ureteral stent design, materials and coatings. Expert Rev Med Devices. 2006 May;3(3):395-403. doi: 10.1586/17434440.3.3.395. PMID 16681460
- [Background] Joshi HB, Newns N, Stainthorpe A, MacDonagh RP, Keeley FX Jr, Timoney AG. Ureteral stent symptom questionnaire: development and validation of a multidimensional quality of life measure. J Urol. 2003 Mar;169(3):1060-4. doi: 10.1097/01.ju.0000049198.53424.1d. PMID 12576846